CLINICAL TRIAL: NCT04803877
Title: SARC038: A Phase 2 Study of Regorafenib in Combination With Nivolumab in Patients With Refractory or Recurrent Osteosarcoma
Brief Title: SARC038: Phase 2 Study of Regorafenib and Nivolumab in Osteosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC038
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Osteosarcoma; Osteosarcoma in Children; Osteosarcoma Recurrent; Osteosarcoma Metastatic
MeSH Terms: conditions — Osteosarcoma | interventions — regorafenib; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib and Nivolumab (Experimental)
  Interventions: Drug: Regorafenib 40 MG; Drug: Regorafenib 20MG; Drug: Nivolumab

INTERVENTIONS:
Drug: Regorafenib 40 MG — For subjects age 18 and older, Regorafenib will be administered as 80mg oral once daily on Cycle 1, Days 1-7 and then escalated to 120 mg once daily for Cycle 1, Days 8-21 if no Grade 2 or above regorafenib adverse events occur. For subsequent cycles, the highest tolerated dose will be taken once daily on days 1-21 of each 28-day cycle.
Drug: Regorafenib 20MG — For subjects younger than 18 years, Regorafenib will be administered as 60mg/m2/dose (rounded to the nearest 20mg, maximum dose of 80mg) once daily for Cycle 1, Days 8-21 if no Grade 2 or above regorafenib-related adverse events occur. For subsequent cycles, the highest tolerated dose will be taken once daily on days 1-21 of each 28-day cycle.
Drug: Nivolumab — For subjects age 18 and older, Nivolumab will be administered at 480mg IV over 30 min every 28 days.
  For subjects younger than 18 years, Nivolumab 3mg/kg (maximum dose 240mg) will be administered IV over 30 minutes on day 1 and 15 of each 28-day cycle.

SUMMARY:
A phase 2 study of regorafenib in combination with nivolumab in patients with refractory or recurrent osteosarcoma.

DETAILED DESCRIPTION:
This is a single arm, Simon two-stage historically controlled study to compare the 4 month progression-free survival rate of patients with relapsed/refractory osteosarcoma treated with regorafenib in combination with nivolumab to those who received regorafenib alone (historical control).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years at the time of enrollment. Every effort will be made to ensure that 50% of patients will be ≤ 21 years of age.
* Histologically confirmed high grade osteosarcoma (excluding osteosarcoma associated with Paget disease of bone or extraskeletal osteosarcoma) at diagnosis or relapse.

Must have relapsed or refractory osteosarcoma following at least one line of systemic therapy for the initial treatment of osteosarcoma.

* Performance Status: Lansky (≤ 16 years of age) or Karnofsky (>16 years of age) performance score of ≥ 70, or Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1. See Appendix A. Patients who are unable to walk because of paralysis, but who are up and about in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* At least one site of measurable disease on CT/MRI scan as defined by RECIST 1.1. Baseline imaging must be performed within 21 days of Day 1 of study therapy.
* Must be able to swallow intact pills
* Adequate organ and bone marrow function within 7 days of Day 1 of study therapy defined as:
* Absolute Neutrophil Count (ANC) ≥ 1000/mm3
* Platelets ≥ 75 000/mm3
* Hemoglobin ≥ 8 g/ dL (transfusions allowed)
* ALT and AST ≤ 3 x institutional upper limit of normal (ULN) or ≤ 5.0 x institutional ULN if considered due to tumor
* Serum albumin ≥ 3 g/dL
* Serum total bilirubin ≤ 1.5 x institutional ULN. NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study
* Serum creatinine ≤ 3 x institutional ULN or 24-hour creatinine clearance ≥ 30 ml/min (calculated creatinine clearance using Cockcroft formula is acceptable)
* Normal free T4. Replacement therapy allowed.
* Serum lipase ≤ 1.5 x ULN
* INR ≤ 1.5 x ULN
* Urine protein: Meets one of the following criteria: (i) urinary protein by urine dipstick is ≤ 100mg/dL or ≤ 2+ (ii) Urine Protein Creatinine(UPC) ratio <3.5 (iii) 24-hour urine protein was measured, urinary protein ≤ 3500 mg
* Adequate pulmonary function defined as:
* No evidence of dyspnea at rest
* No activity limitation due to pulmonary insufficiency
* Pulse Oximetry >92% on room air
* Adequate cardiac function defined as:
* QTc ≤ 480 msec
* Shortening fraction ≥ 27% by echocardiogram or ejection fraction ≥ 50% by gated radionuclide study or echocardiogram
* No congestive heart failure (CHF) worse than New York Heart Association Functional Classification Class I.
* No clinically significant cardiac arrhythmias, stroke or myocardial infarction within 6 months prior to enrollment.
* Prior Therapy: All prior treatment-related toxicities must have resolved to ≤ Grade 1 or be determined clinically stable by the Investigator.
* Myelosuppressive chemotherapy: Patients must not have received myelosuppressive chemotherapy within 3 weeks of enrollment
* Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a white blood cell or platelet growth factor. At least 14 days must have elapsed after receiving pegfilgrastim.
* Biologic (anti-neoplastic agent): At least 7 days must have elapsed since completion of therapy with a biologic agent.
* Monoclonal antibodies: At least 21 days must have elapsed since prior therapy that included a monoclonal antibody (e.g., dinutuximab, denosumab, bevacizumab).
* Radiotherapy: ≥ 2 weeks must have elapsed since local palliative XRT (small port); ≥ 3 months must have elapsed if prior craniospinal XRT was received, if ≥ 50% of the pelvis was irradiated, or if TBI was received; ≥ 6 weeks must have elapsed if other substantial bone marrow irradiation was given.
* Autologous Stem Cell Transplant or Rescue or Cellular Therapy: ≥ 2 months must have elapsed since transplant/cellular therapy.
* Voluntary, written informed consent
* Negative urine or serum pregnancy test in women of childbearing potential. Women of childbearing potential includes pre-menarchal girls with evidence of puberty onset, and adult women through the end of the first 2 years of the onset of menopause. Testing should be completed ≤ 7 days prior to Day 1 of study.
* Fertile men and women of childbearing potential must agree to use an effective method of birth control from Day 1 of study and for 5 months after last dose of nivolumab or for 8 weeks after last dose of regorafenib, whichever is longer.
* Effective methods of birth control include: surgical sterility (subject or subject's partner), barrier device (condom, diaphragm), contraceptive coil (IUD), abstinence, or oral contraception.
* Patients with central nervous system (CNS) disease are eligible if they have received prior radiotherapy or surgery to sites of CNS metastatic disease and are without evidence of progression for at least 4 weeks after CNS therapy.

Patients >18 years must be willing to undergo tumor biopsy at study entry and post-treatment biopsy for biologic correlates. If biopsy is contra-indicated, enrollment must be approved by study PI and archival tissue must be available.

Exclusion Criteria:

* Patients with prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen in this trial.
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery (thoracotomy or laparotomy, etc.), laparoscopic biopsy, or significant traumatic injury within 28 days prior to Day 1 of study or who have not recovered adequately from prior surgery
* Women who are pregnant or nursing/breastfeeding.
* Known hypersensitivity to excipients of the formulations of regorafenib or nivolumab or similar agents
* Inability to comply with protocol required procedures
* Prior therapy with an immune checkpoint inhibitor or a tyrosine kinase inhibitor targeting VEGF
* Patients with autoimmune disease.
* Chronic use of immunosuppressive therapies
* Received any investigational drug within 28 days of study enrollment
* Uncontrolled infection
* Known active HIV. Testing is not required. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. However, strong CYP3A4 inhibitors are prohibited.
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Prior allogeneic hematopoietic stem cell/bone marrow transplant or solid organ transplant
* Uncontrolled hypertension defined as on average, > 140 systolic pressure or > 90 diastolic pressure in patient ≥ 18 y/o or > 95th percentile for age/gender in patients < 18 y/o despite medical management. If blood pressure is borderline, ensure patient is properly prepared (relaxed, sitting in chair for > 3 minutes), proper technique is used (correct cuff size and positioning), and document 2 separate recordings, each at least >5 minutes apart.
* History of clinically significant venous or arterial thrombotic or embolic event requiring systemic anticoagulation within 6 months of enrollment.
* Requirement of oral anticoagulant therapy with oral vitamin K antagonists (warfarin). Low-dose anticoagulants for maintenance of patency of central venous device or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin or direct oral anticoagulants is allowed, providing the event prompting treatment occurred > 6 months prior. Subjects who are prophylactically being treated with an agent such as heparin will be allowed to participate, provided no prior evidence of underlying abnormality in coagulation parameters exists.
* Presence of non-healing wound, non-healing ulcer or fracture (excluding pathologic fracture)
* Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE Grade 2 dyspnea)
* Significant currently active gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, malabsorption, or CTCAE Grade ≥ 2 diarrhea of any etiology
* Patients with history of bowel perforation or fistula formation.
* Live/attenuated vaccine administered within 30 days of enrollment
* Patients receiving or requiring strong CYP3A4 inhibitors (e.g., clarithromycin, grapefruit juice, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifampin, St. John's wort)
* Any hemorrhage or bleeding event CTCAE ≥ Grade 3 within 28 days of study enrollment
* Body surface area (BSA) < 0.4 m2

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Compare the 4-month progression-free survival rate to historical controls | Approximately 4 months
  To compare the 4-month progression-free survival (PFS) rate in patients with relapsed or refractory osteosarcoma administered regorafenib in combination with nivolumab to historical controls who received regorafenib alone, as per iRECIST. PFS will be determined as the time from the start of study treatment (Cycle 1, Day 1) to time of disease relapse, disease progression, or death from any cause, using iRECIST. The proportion of patients who do not experience one of these events at 4 months will be determined.

SECONDARY OUTCOMES:
Objective Response Rate | Approximately 5 years
  To estimate the objective response rate (ORR) in patients with relapsed or refractory osteosarcoma administered regorafenib in combination with nivolumab, according to iRECIST. Objective tumor response, defined as achievement of nadir response of complete response (CR) or partial response (PR) by iRECIST without prior progression any time during protocol therapy.
Progression-Free Survival | Approximately 5 years
  To estimate the PFS, including median PFS, in this population. Progression-free survival (PFS) defined as the time from study entry to disease relapse, disease progression, or death from any cause, using iRECIST. Patients without an event will be censored at the time of last disease follow-up.
Progression-Free Survival and Objective Response Rate | Approximately 5 years
  To compare the 4-month PFS rate and ORR to historical controls in this population, according to RECIST 1.1. Duration of response is defined as the time from a nadir tumor response of CR/PR to disease progression.
Describe adverse events | Approximately 5 years
  To describe the toxicities of regorafenib in combination with nivolumab in patients with relapsed or refractory osteosarcoma. Adverse events will be graded as defined in CTCAE v. 5.0 during each therapy course.
Estimate 1-year and 2-year Overall Survival | Approximately 5 years
  To estimate 1-year and 2-year overall survival (OS) in patients with relapsed or refractory osteosarcoma treated with regorafenib in combination with nivolumab. Overall survival, defined as the time from study entry to death from any cause. Patients who are alive at the time of analysis will be censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Miami, Miami, Florida
  - Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's, Cincinnati, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas